CLINICAL TRIAL: NCT01409707
Title: Mechanisms of Change, Motivation, and Treatment Outcome in AD-PTSD
Brief Title: Mechanisms of Change, Motivation, and Treatment Outcome in Alcohol Dependence - Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Scott F. Coffey, Professor and Director, Division of Psychology, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-0071; R01AA016816 (NIH)
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-01

CONDITIONS: Alcohol Dependence; Posttraumatic Stress Disorder
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy lifestyles sessions (Experimental): Healthy lifestyles sessions is a structured 9-12 session intervention that provides education about a variety of health-related topics. Each therapy session was 50-60 minutes long. Sessions included the provision of information, discussing participants' understanding of information, and answering questions about the information provided.
  Interventions: Behavioral: Healthy lifestyles sessions
- Trauma-focused exposure therapy (Experimental): Trauma focused exposure therapy is a well-described cognitive-behavioral therapy that utilizes imaginal and in vivo exposure techniques to reduce the symptoms of posttraumatic stress disorder. In addition to imaginal and iv vivo exposure techniques, in the current study patients were provided psychoeducation about posttraumatic stress disorder, a rationale for trauma focused exposure therapy, and were taught breathing retraining as a method to manage arousal associated with posttraumatic stress disorder. Nine to 12 50-60 minutes sessions were provided.
  Interventions: Behavioral: Trauma-focused exposure therapy
- Motivational enhancement + trauma-focused exposure therapy (Experimental): A one session, 90 min. trauma-focused motivational enhancement therapy session was provided prior to starting the trauma-focused exposure therapy. Trauma focused exposure therapy is a well-described cognitive-behavioral therapy that utilizes imaginal and in vivo exposure techniques to reduce the symptoms of posttraumatic stress disorder. In addition to imaginal and iv vivo exposure techniques, in the current study patients were provided psychoeducation about posttraumatic stress disorder, a rationale for trauma focused exposure therapy, and were taught breathing retraining as a method to manage arousal associated with posttraumatic stress disorder. Nine to 12 50-60 minutes sessions were provided.
  Interventions: Behavioral: Motivational enhancement + trauma-focused exposure therapy

INTERVENTIONS:
Behavioral: Trauma-focused exposure therapy — cognitive behavioral therapy for PTSD
  Other Names: Prolonged exposure
  Arms: Trauma-focused exposure therapy
Behavioral: Motivational enhancement + trauma-focused exposure therapy — Cognitive behavioral therapy for PTSD
  Other Names: Trauma-focused motivational enhancement therapy; Prolonged Exposure; Motivational Interviewing
  Arms: Motivational enhancement + trauma-focused exposure therapy
Behavioral: Healthy lifestyles sessions
  Arms: Healthy lifestyles sessions

SUMMARY:
The purpose of this study is to test if provision of an effective psychotherapy for Post-traumatic Stress Disorder (PTSD), prolonged exposure, can be tolerated in alcohol dependent patients with PTSD and if it is associated with better treatment outcomes compared to an active control condition.

ELIGIBILITY:
Inclusion Criteria:

* Current PTSD
* Current Alcohol Dependence
* at least one heavy drinking day in the past 60 days

Exclusion Criteria:

* Psychotic disorder
* Untreated bi-polar disorder
* benzodiazepine use

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2008-07; Primary Completion 2012-01 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott F. Coffey, Ph.D., Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at a residential substance abuse treatment facility between July 2008 and June 2011.
Pre-assignment Details: 222 assessed; 96 ineligible. 53 did not have current PTSD, 6 did not have current alcohol dependence (AD), and 2 did not have either current PTSD or AD. 35 participants were ineligible for other reasons (e.g., current mania, current psychosis, etc.).
Groups:
- Trauma-focused Exposure Therapy: Trauma-focused exposure therapy is a well-described cognitive-behavioral therapy that utilizes imaginal and in vivo exposure techniques to reduce the symptoms of posttraumatic stress disorder. In addition to imaginal and iv vivo exposure techniques, in the current study patients were provided psychoeducation about posttraumatic stress disorder, a rationale for trauma-focused exposure therapy, and were taught breathing retraining as a method to manage arousal associated with PTSD. Nine to 12 50-60 minutes sessions were provided.
- Motivational Enhancement + Trauma-focused Exposure Therapy: A one session, 90 min. trauma-focused motivational enhancement therapy session was provided prior to starting exposure therapy. Exposure therapy is a well-described cognitive-behavioral therapy that utilizes imaginal and in vivo exposure techniques to reduce the symptoms of posttraumatic stress disorder. In addition to imaginal and iv vivo exposure techniques, in the current study patients were provided psychoeducation about posttraumatic stress disorder, a rationale for exposure therapy, and were taught breathing retraining as a method to manage arousal associated with posttraumatic stress disorder. Nine to 12 50-60 minutes sessions were provided.
Period: Overall Study
Arm/Group | Healthy Lifestyles Sessions | Trauma-focused Exposure Therapy | Motivational Enhancement + Trauma-focused Exposure Therapy
Started | 41 | 45 | 40
Completed | 36 | 28 | 24
Not Completed | 5 | 17 | 16
Not completed — Withdrawal by Subject | 5 | 17 | 16

BASELINE CHARACTERISTICS:
Groups:
- Healthy Lifestyles Sessions: HLS is a structured 9-12 session intervention that provides education about a variety of health-related topics. Each therapy session was 50-60 minutes long. Sessions included the provision of information, discussing participants' understanding of information, and answering questions about the information provided.
- Trauma-focused Exposure Therapy: EXP is a well-described cognitive-behavioral therapy that utilizes imaginal and in vivo exposure techniques to reduce the symptoms of PTSD. In addition to imaginal and iv vivo exposure techniques, in the current study patients were provided psychoeducation about PTSD, a rationale for EXP, and were taught breathing retraining as a method to manage arousal associated with PTSD. Nine to 12 50-60 minutes sessions were provided.
- Motivational Enhancement + Trauma-focused Exposure Therapy: A one session, 90 min. trauma-focused motivational enhancement therapy session was provided prior to starting the trauma-focused exposure therapy. EXP is a well-described cognitive-behavioral therapy that utilizes imaginal and in vivo exposure techniques to reduce the symptoms of PTSD. In addition to imaginal and iv vivo exposure techniques, in the current study patients were provided psychoeducation about PTSD, a rationale for EXP, and were taught breathing retraining as a method to manage arousal associated with PTSD. Nine to 12 50-60 minutes sessions were provided.
- Total: Total of all reporting groups
Arm/Group | Healthy Lifestyles Sessions | Trauma-focused Exposure Therapy | Motivational Enhancement + Trauma-focused Exposure Therapy | Total
Number analyzed (Participants) | 41 | 45 | 40 | 126
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 41 | 45 | 40 | 126
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.85 (10.67) | 34.67 (10.33) | 34.40 (10.65) | 33.72 (10.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 18 | 58
  Male | 20 | 26 | 22 | 68
Region of Enrollment [Number; unit: participants]
  United States | 41 | 45 | 40 | 126

OUTCOME MEASURES:

1. Primary Outcome: Impact of Event Scale-Revised
Description: The Impact of Event Scale-Revised is a 22-item self-report measure of posttraumatic stress disorder symptoms. The total score for the Impact of Event Scale-Revised ranges from 0 to 88 with lower scores representing less severe symptoms of posttraumatic stress disorder and higher scores representing more severe symptoms of posttraumatic stress disorder.
Time Frame: 3-months posttreatment
Population: All participants who started the study were included in the analyses (ITT). Missing data were estimated using maximum likelihood estimation.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Motivational Enhancement + Trauma-focused Exposure Therapy: One 90 min. motivational enhancement therapy session was provided prior to beginning trauma focused therapy. EXP is a well-described cognitive-behavioral therapy that utilizes imaginal and in vivo exposure techniques to reduce the symptoms of PTSD. In addition to imaginal and iv vivo exposure techniques, in the current study patients were provided psychoeducation about PTSD, a rationale for EXP, and were taught breathing retraining as a method to manage arousal associated with PTSD. Nine to 12 50-60 minutes sessions were provided.
Arm/Group | Healthy Lifestyles Sessions | Trauma-focused Exposure Therapy | Motivational Enhancement + Trauma-focused Exposure Therapy
Number analyzed (Participants) | 41 | 45 | 40
units on a scale | 26.00 (2.98) | 19.10 (3.10) | 14.11 (2.95)
Statistical Analysis 1: Comparison: Healthy Lifestyles Sessions vs Trauma-focused Exposure Therapy vs Motivational Enhancement + Trauma-focused Exposure Therapy; Multilevel mixed modeling was employed. The null hypothesis was that there'd be no differences between groups at posttreatment on posttraumatic stress disorder measures or alcohol use measures; Test type: Superiority or Other; p = .068, Mixed Models Analysis — The a priori threshold for statistical significance was set at p = .05

2. Primary Outcome: Timeline Follow Back
Description: The timeline follow back is a measure of drug and alcohol consumption in the prior 90 days. The timeline follow back is a calendar-based retrospective account of drug and alcohol consumption for a specified period of time (e.g., past 90 days). One of the most commonly reported metrics of drug and alcohol consumption from this measure is percent days abstinent (PDA). Percent days abstinent is simply the proportion of days for the specified period of time (e.g., 90 days) in which drugs or alcohol were not consumed. Percent days abstinent can range from 0 to 100 with 0 representing no abstinence during a specified period of time (i.e., consumed alcohol every day) and 100 representing complete abstinence during a specified period of time.
Time Frame: 3-months posttreatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of days abstinent
Arm/Group | Healthy Lifestyles Sessions | Trauma-focused Exposure Therapy | Motivational Enhancement + Trauma-focused Exposure Therapy
Number analyzed (Participants) | 41 | 45 | 40
percentage of days abstinent | 97.95 (4.25) | 97.83 (4.30) | 92.12 (4.38)
Statistical Analysis 1: Comparison: Healthy Lifestyles Sessions vs Trauma-focused Exposure Therapy vs Motivational Enhancement + Trauma-focused Exposure Therapy; Multilevel mixed modeling was employed. The null hypothesis was that there would be no differences in alcohol use at posttreatment; Test type: Superiority or Other; p = 0.39, Mixed Models Analysis — The a priori threshold for statistical significance was set at p=.05

ADVERSE EVENTS:
Arm/Group | Healthy Lifestyles Sessions | Trauma-focused Exposure Therapy
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/82
Other Adverse Events (participants affected / at risk) | 0/38 | 0/82

LIMITATIONS AND CAVEATS:
Unclear whether results will generalize to outpatient sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No